CLINICAL TRIAL: NCT05898308
Title: Comparison of a Personalized Maintenance Therapy Based on the Evolution of Anti-desmoglein Antibodies as Biomarkers of Pemphigus Subclinical Activity, With the Standard Treatment (Rituximab + Corticosteroids) in Pemphigus
Brief Title: Comparison of a Personalized Maintenance Therapy With the Standard Treatment in Pemphigus
Acronym: RITUX4
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/0424/HP
Record Dates: First submitted 2023-05-26; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Pemphigus; Dermatologic Disease
Keywords: Pemphigus; Rituximab; Biomarkers; Personalized medicine
MeSH Terms: conditions — Pemphigus; Skin Diseases | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: In both arms, patients will be initially treated according to the French guidelines (PNDS) based on the Ritux-3 regimen: 1000 mg of rituximab on Day1-Day14, and 500 mg at Month 12 and Month 18, plus oral prednisone 1 mg/kg/day initially, with the aim to stop prednisone after 6 months.
  "standard-of-care" arm will be treated as mentioned above. "personalized maintenance treatment" arm will be treated with the same regimen, adapted according to the evolution of anti-Dsg Abs: During the initial phase of treatment: patients i) whose serum anti-Dsg Abs have not sufficiently decreased ii) and/or those who initially had a severe pemphigus (at the inclusion visit) defined by a PDAI score > 45) will receive 1 g of rituximab at Month 6 ; the second year from Month 22 (4 months after the Month 18 infusion of 500 mg of rituximab) until the end of the study: patients whose anti-Dsg3 Abs re-increase >50 UI/ml and/or anti-Dsg1Abs re-increase>20 UI/ml) will receive 1 g of rituximab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "standard-of-care" arm (No Intervention): Patients will be initially treated according to the French guidelines (PNDS) based on the Ritux-3 regimen: 1000 mg of rituximab on Day1-Day14, and 500 mg at Month 12 and Month 18, plus oral prednisone 1 mg/kg/day initially, with the aim to stop prednisone after 6 months.
  The prednisone dose could be increased up to 1.5 mg/kg/day in patients who do not achieve disease control with the initial 1 mg/kg/day dose.
- "personalized maintenance treatment" arm (Experimental): Patients will be treated with the same regimen (1000 mg of rituximab on Day1-Day14, and 500 mg at Month 12 and Month 18, plus oral prednisone 1 mg/kg/day initially, with the aim to stop prednisone after 6 months), which will then be adapted according to the evolution of anti-Dsg Abs: During the initial phase of treatment: patients i) whose serum anti-Dsg Abs have not sufficiently decreased ii) and/or those who initially had a severe pemphigus (at the inclusion visit) defined by a PDAI score > 45) will receive 1 g of rituximab at Month 6 ; Beyond the second year from Month 22 (4 months after the Month 18 infusion of 500 mg of rituximab) until the end of the study: patients whose anti-Dsg3 Abs re-increase >50 UI/ml and/or anti-Dsg1Abs re-increase>20 UI/ml) will receive 1 g of rituximab. A maximum of 2 additional maintenance infusions of rituximab per year will be allowed during the study.
  Interventions: Drug: RiTUXimab Injection

INTERVENTIONS:
Drug: RiTUXimab Injection — Patients assigned to the "personalized maintenance treatment" will be treated by additional RITUXIMAB injection depending on anti-Dsg Abs levels.
  Arms: "personalized maintenance treatment" arm

SUMMARY:
Pemphigus diseases are life-threatening chronic autoimmune blistering diseases characterized by split formation within the epidermis and surface-close epithelia accompanied by acantholysis. Autoantibodies (Abs) are mainly directed against two structural proteins of the epidermal/epithelial desmosome, desmoglein (Dsg) 1 and Dsg3. Two main pemphigus variants can be differentiated, pemphigus vulgaris (PV), and pemphigus foliaceus (PF). Diagnosis of PV and PF is based on the combination of the clinical picture, histological picture of acantholysis, direct immunofluorescence microscopy (DIF) of a perilesional biopsy and serology.

The present "Ritux 4" trial is the fourth academic study with the French study group on auto immune bullous skin diseases (Groupe Bulle) to assess the use of rituximab in auto immune bullous skin diseases, in particular pemphigus. The 3 previous trials have been published in outstanding Journals (N Engl J Med 2007, Science Transl Med 2013, The Lancet 2017 and 2020), and have led to the approval of rituximab in pemphigus by the FDA in 2018 and EMA in 2019. In addition, an industry-sponsored trial testing rituximab versus mycophenolate mofetil in pemphigus, that the investigators have largely contributed to design has been very recently accepted for publication in the N Engl J Med (2021).

The investigator hypothesize that a maintenance therapy using an infusion of 1g of rituximab at Month 6 in patients whose anti-Dsg Abs have not sufficiently decreased at Month 3 after the initial cycle of rituximab (persistence of anti-Dsg1 Abs> 20 UI/ml and/or anti-Dsg3 Abs> 130 UI/ml), and or had an initial PDAI score >45 ( first year of follow-up), and the re-treatment with 1g of rituximab of patients whose anti Dsg Abs re-increase during the evolution of pemphigus after the initial cycle of rituximab (anti-Dsg1 Abs> 20 IU/ml, anti-Dsg3 Abs> 50 UI/ml), could be effective in preventing the occurrence of relapses, thus avoiding to restart a CS treatment, and would provide benefit as compared with the current treatment strategy of retreating patients with 2 g of rituximab (1g at Day0 and Day14) combined with oral CS patients, once a clinical relapse occurs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years
* Signed Informed Consent Form (or from the family in case of impossibility of patient's consent).
* Confirmed newly diagnosed PV or PF, based on the presence of the following: histological features of acantholysis on skin or mucosal biopsy, and deposition of IgG, complement component 3, or both on the keratinocyte membrane detected by direct immunofluorescence on affected skin or mucosa
* Presence of moderate-to-severely active disease, defined by an overall PDAI score> 1554
* Patient able to receive the standard-of-care consisting of corticosteroids (prednisone 1 mg/kg/day PO) and rituximab
* Patients must be vaccinated against Covid-19 before study entry. It is recommended that patients are vaccinated against influenza and Streptococcus pneumoniae and have their first injection (Prevenar 13) before study entry.
* For women who are not postmenopausal (menopausal: ≥ 12 months of non-therapy-induced amenorrhoea) or surgically sterile (absence of ovaries and/or uterus + bilateral salphingectomy) and who do not plan on having children anymore: agreement to remain abstinent or use two adequate methods of contraception, including at least one method with a failure rate of <1% per year, during the treatment period and for at least 12 months after the last dose of study treatment. They must have a negative result from a blood beta-HCG test within 1 week prior to randomization Abstinence is acceptable only if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Barrier methods must always be supplemented with the use of a spermicide.

• For men: Surgical sterility or agreement to remain abstinent or use a condom during the treatment period and for at least 12 months after the last dose of study treatment and agreement to refrain from donating sperm during this same period.

Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient.

Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

* Able to comply with the study protocol, in the investigator's judgment
* Patient affiliated with, or beneficiary of a social security (national health insurance) plan

Exclusion Criteria:

* Non-consenting patient or patient who cannot be followed regularly.
* Diagnosis of paraneoplastic pemphigus or evidence of other non-PV or PF autoimmune blistering disease
* Contraindication to rituximab marketed as 500 mg concentrate for solution for infusion
* Contraindication to prednisone marketed as 20 mg, scored tablet pharmaceutical form
* Contraindication to methylprednisolone marketed as 120 mg powder for injectable solution pharmaceutical form
* Contraindication to paracetamol marketed as 10 mg/mL solution for infusion pharmaceutical form
* Contraindication to dexchlorpheniramine maleate marketed as 5 mg/1mL injectable solution pharmaceutical form
* Lack of peripheral venous access
* Pregnant or lactating
* Significant cardiovascular or pulmonary disease (including obstructive pulmonary disease)
* Evidence of any new or uncontrolled concomitant disease that, in the investigator's judgment, would preclude patient participation, including but not limited to nervous system, renal, hepatic, endocrine, malignant, or gastrointestinal disorders
* Any concomitant condition that required treatment with oral or systemic corticosteroids within 12 weeks prior to randomization- excluding transitory treatments (such as a corticosteroid therapy prescribed for a few days for an acute infection), and chronic corticosteroid treatments with a prednisone / prednisolone dose ≤20 mg/day, (these latter patients remain eligible for study entry)
* Treatment with IV Ig, plasmapheresis, or other similar procedure within 8 weeks prior to randomization
* Patients having received immunosuppressive treatment (such as cyclosporine, mycophenolate mofetil, azathioprine given at an effective dose for any other condition than Pemphigus, or any other treatment that might potentially be active on Pemphigus lesions (anti-TNF) within 4 weeks prior to baseline
* Treatment with cyclophosphamide within 12 weeks prior to randomization
* Patients with positive blood test for HIV
* Inherited or acquired severe immune deficiency
* Known active infection of any kind (excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV anti-infectives within 4 weeks prior to screening, or completion of oral anti-infectives within 2 weeks prior to randomization. Entry into this study may be reconsidered once the infection has fully resolved.
* Patients with a currently treated cancer, including solid tumors, hematologic malignancies, and carcinoma (except basal cell of the skin and squamous cell carcinoma of the skin which can be easily cured with a standard excision )
* Patients with a past history ( < 5 years) of cancer, including solid tumors, hematologic malignancies, and carcinoma (except complete excision of basal cell of the skin and squamous cell carcinoma of the skin that have been excised and cured) NB: Patients whose cancer is cured and do not have anti-cancer treatment anymore must be referred to an oncologist before entry in the study
* Currently active alcohol or drug abuse, or history of alcohol or drug abuse within 24 weeks prior to screening
* Major surgery within 4 weeks prior to randomization, excluding diagnostic surgery
* Treatment with rituximab or a B cell-targeted therapy (e.g., anti-CD20, anti-CD22, or anti-BLyS) within 12 months prior to randomization
* Treatment with a live or attenuated vaccine within 28 days prior to randomization. It is recommended that a patient's vaccination record and the need for immunization prior to study entry be carefully investigated.
* Major biological abnormality which in the investigator's judgment, would preclude patient participation,
* Positive test results for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus (HCV) serology at screening
* Participation in another interventional clinical trial within 28 days prior to randomization and during the study
* Person deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of relapses/ flares by patient-year, defined according to the pemphigus consensus statement | 7.5 years
  by the appearance of 3 or more new lesions a month that do not heal spontaneously within 1 week, or by the extension of established lesions, in a patient who has achieved disease control.
  Unit : /patient/year

SECONDARY OUTCOMES:
Number of patients-years of additional rituximab infusions to avoid one relapse by year (Number needed to treat, NNT). | 7.5 years
  Unit: none (ratio of variables with the same dimension)
Time to disease flare/ relapse | 7.5 years
  Unit : years
Cumulative duration of complete remission during the study | 7.5 years
  Unit : % of the time
Number of maintenance infusions of 2 g of rituximab per patient-year | 7.5 years
  Unit: /patient/year
Cumulative dose of rituximab by patient-year | 7.5 years
  Unit : g/patient/year
blood leukocytes (measured at D15, M1, then every 3 month from M3 to M48) | 7.5 years
  Unit : count/mL
anti-Dsg1 IgG measured by ELISA (measured at D15, M1, M2, then every 3 month from M3 to M48) | 7.5 years
  Unit : UI/mL
anti-Dsg3 IgG measured by ELISA (measured at D15, M1, M2, then every 3 month from M3 to M48 | 7.5 years
  Unit : UI/mL
Quality of life, using the French version of bullous specific QOL questionnaire | 7.5 years
  Measured at M1, M2, every 3 months from M3 to M48, averaged on all follow-up visits (area under curve) Unit : ABQOL/TABQOL points

CONTACTS AND LOCATIONS:
Overall Officials: Pascal JOLY, Principal Investigator — University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No